CLINICAL TRIAL: NCT03652896
Title: Anatomy-based Resection or Margin-based Resection for Hepatocellular Carcinoma: A Randomized Controlled Trial
Brief Title: Anatomy-based Resection or Margin-based Resection for Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaoping Chen, Professor and Chairman, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AR2018MR
Record Dates: First submitted 2018-08-20; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Hepatocellular Carcinoma by BCLC Stage
Keywords: hepatocellular carcinoma; anatomical liver resection
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anatomical liver resection (Experimental): resect the tumor located liver segment or lobe
  Interventions: Procedure: anatomical liver resection
- resection margin based liver resection (Experimental): non-anatomical liver resection, but insure adequate resection margin
  Interventions: Procedure: anatomical liver resection

INTERVENTIONS:
Procedure: anatomical liver resection — Liver resection is performed to achieve R0 resection for patients with appropriate BCLC staging, indocyanine green retention rate, Child-pugh grading and adequate liver remnant.
  Other Names: non-anatomical liver resection

SUMMARY:
Anatomical liver resection was widely accepted as first line curative therapy for hepatocellular carcinoma. However, number of retrospective clinical studies showed no priority of anatomical resection for hepatocellular, compared with non-anatomical resection.

Surgical resection margin is a essential factor that may affect tumor prognosis. It is controversial whether adequate liver resection margin is associated with improved survival outcome in patients with hepatocellular.

There was few prospective clinical trial to investigate whether anatomical liver resection is superior to non-anatomical resection or liver resection with adequate margin is superior to that with inadequate margin. This prospective clinical trial aims at fix these issues.

DETAILED DESCRIPTION:
In the anatomical liver resection group, liver segmentectomy or lobectomy is performed to insure curative resection (R0 resection). The region of liver resected is based on the anatomy or portal vein and hepatic vein. The liver pedicle of the tumor located lobe is exposed and dissected, which is principle to perform anatomical liver resection.

In the non-anatomical liver resection group, the liver parenchyma transection is around 0-2 cm from the tumor margin, according to tumor size and location.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with hepatocellular carcinoma of BCLC stage A
* liver function Child-pugh A
* normal indocyanine green retention rate
* adequate liver remnant

Exclusion Criteria:

* age less than 17 y or older than 65 y
* unresectable liver cancer
* intraoperative ablation
* contraindication for liver resection
* preoperative treatment for hepatocellular
* active hepatitis
* pregnant
* multi-original tumors
* mixed liver cancer (hepatocellular carcinoma and cholangiocellular carcinoma)
* tumor recurrence

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
prognosis | 5 years
  3 year and 5 year overall survival and disease free survival

SECONDARY OUTCOMES:
postoperative recovery | 30 days postoperatively
  postoperative complications
hospital stay | 60 days postoperatively
  hospital days after operation

OTHER OUTCOMES:
surgery duration | 24 hours
  time duration of liver parenchyma transection
volume of bleeding | 24 hours
  millilitre of blood lost during operation
volume of transfusion | 24 hours
  units of blood transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Chen, M.D., Principal Investigator — Huazhong University of Science and Technology
Locations (1):
- Hepatic Surgery Center of Tongji Hospital, Wuhan, Hubei, China